CLINICAL TRIAL: NCT06568926
Title: Adherence of Beta Thalssemia Patients to Oral Chelation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Aly Mousa, Resident-pediatric department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med-24-07-17MS
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient group (Experimental): Beta thalassemia patients on oral chelation therapy
  Interventions: Diagnostic Test: Serum Ferritin level

INTERVENTIONS:
Diagnostic Test: Serum Ferritin level — follow up to the ferritin level in beta thalaseemia patients on oral chelation therapy

SUMMARY:
The β-thalassemias are a group of inherited disorders of hemoglobin (Hb) synthesis characterized by chronic anemia of varying severity. The degree of anemia relies on several genetic and environmental factors and determines the need for regular transfusion therapy. It is now common practice to classify patients as having transfusion dependent β-thalassemia (TDT) or non-transfusion-dependent β-thalassemia (NTDT). Regarding geographical distribution of β-thalassemia, it prevails more in countries on the Mediterranean, South east of Asia and in the east of Europe. In Egypt, it is the most common cause of chronic blood loss: One thousand cases are recorded annually for every 1.5 million live births the disease prevalence is equal to1000 cases per 1.5 million live births (Ghazala et al., 2021).

The only curative treatment for thalassemia currently is a bone marrow transplant. However, it is restricted to only a few patients due to the non-availability of an HLA-matched donor and high cost. Thus, most patients receive regular blood transfusions accompanied by iron chelation therapy (ICT) as the standard of care. The ideal management of a patient with transfusion-dependent thalassemia (TDT) requires a multidisciplinary therapeutic approach. The main iron chelating agents include deferoxamine (DFO), deferiprone (DFP), and deferasirox (DFX). Due to poor oral bioavailibility, DFO is the only chelator that must be administered subcutaneously or intravenously up to once a day; DFP and DFX may be administered orally up to three times a day. The known side effects associated with each chelator include infusion reactions in DFO, gastrointestinal distress, agranulocytosis in DFP, and transaminitis in DFP and DFX.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of beta thalassemia major or intermedia,
2. Age between 2-18 years,
3. Receiving regular blood transfusions every 2-5 weeks
4. Prescribed oral iron chelation therapy with deferasirox for at least 1 year prior to enrollment.

Exclusion Criteria:

1. Age less than 2 years and more than 18 years
2. Any cause of blood transfusion other than beta Thalassemia
3. Patients on deferoxamine

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
serum ferritin level in beta thalassemia patients adherent to oral chelation therapy | 1 year
  Adherence of Beta Thalssemia Patients to Oral Chelation Therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belhoul KM, Bakir ML, Saned MS, Kadhim AM, Musallam KM, Taher AT. Serum ferritin levels and endocrinopathy in medically treated patients with beta thalassemia major. Ann Hematol. 2012 Jul;91(7):1107-14. doi: 10.1007/s00277-012-1412-7. Epub 2012 Jan 28. PMID 22281991
- [Background] Delea TE, Edelsberg J, Sofrygin O, Thomas SK, Baladi JF, Phatak PD, Coates TD. Consequences and costs of noncompliance with iron chelation therapy in patients with transfusion-dependent thalassemia: a literature review. Transfusion. 2007 Oct;47(10):1919-29. doi: 10.1111/j.1537-2995.2007.01416.x. PMID 17880620
- [Background] Kannan S, Singh A. Compliance score as a monitoring tool to promote treatment adherence in children with thalassemia major for improved physical growth. Asian J Transfus Sci. 2017 Jul-Dec;11(2):108-114. doi: 10.4103/ajts.AJTS_61_16. PMID 28970676
- [Background] Nazir HF, Alshizawi M. Neutropenia and Life-threatening Agranulocytosis Among Children With beta-Thalassemia Treated With Oral Iron Chelators in a Community With Background of Ethnic Neutropenia. J Pediatr Hematol Oncol. 2020 Nov;42(8):e750-e755. doi: 10.1097/MPH.0000000000001699. PMID 31876777